CLINICAL TRIAL: NCT03306823
Title: Multi-center, Single-blind, Prospective Cohort Study of Exploration of Anticoagulation Program in Cerebral Aneurysm and Arteriovenous Malformations With Hybrid Operation
Brief Title: Exploration of Anticoagulation Program in Cerebral Aneurysm and Arteriovenous Malformations With Hybrid Operation 1
Acronym: EAPCAAMHO1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Tang-Du Hospital (Other); Kunming Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other); Nanjing PLA General Hospital (Other); Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Dr. Yong Cao, Principal, Beijing Tiantan Hospital
Other Study IDs: 2016YFC1301800-Anticoagulation
Record Dates: First submitted 2017-05-31; First posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Cerebral Aneurysm; Arteriovenous Malformations
Keywords: Cerebral Aneurysm; Arteriovenous Malformations; Hybrid operation; Anticoagulation
MeSH Terms: conditions — Intracranial Aneurysm; Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- aneurysm: For cerebral aneurysm with hybrid operation, anticoagulation program is decided by different surgeons based on their experience and record the patient's intraoperative activated coagulation time changes in detail.
- arteriovenous malformations: For arteriovenous malformations with hybrid operation, anticoagulation program is decided by different surgeons based on their experience and record the patient's intraoperative activated coagulation time changes in detail.

SUMMARY:
In the stage of registration study, our purpose is to find out the safety range of activated coagulation time level in cerebral aneurysm and arteriovenous malformations with hybrid operation.

DETAILED DESCRIPTION:
This study is divided into anticoagulation program in cerebral aneurysm with hybrid operation and anticoagulation program in cerebral arteriovenous malformations with hybrid operation two parts, and each part divide into two stage, on the stage of registration study. This study is a multi-center, single-blind, prospective cohort study. Record the patient's intraoperative activated coagulation time Changes in detail, to observe the effect of activated coagulation time maintenance level on hemorrhage event rate of Intraoperative and postoperative 48 hours, purpose to find out the safety range of activated coagulation time level in cerebral aneurysm and arteriovenous malformations with hybrid operation. On the stage of randomized controlled study. This study is a multicenter, single-blind, prospective, randomized controlled study. Patients is divided into intraoperative standard dose group of Heparin Sodium and low dose group of Heparin Sodium randomly. To observe the effect of different anticoagulation regimens on activated coagulation time safety coverage rate during surgery, and finally develop a scientific and effective intraoperative anticoagulant therapy program.

ELIGIBILITY:
Inclusion Criteria:

1.All patients undergoing hybird surgery.

Exclusion Criteria:

1. Poor general condition , severe primary disease, surgical contraindications
2. Patient or family refused surgery
3. Fusiform aneurysm,Traumatic aneurysm,Infectious aneurysms
4. Combined with other hemorrhagic cerebrovascular disease
5. Combined with malignant brain tumor
6. Perinatal, Pregnancy
7. Patients unwilling to participate in the trial

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators chose the patiens from the Tiantan hospital and other hospitals that participated in this study.The patients diagnosed as cerebral aneurysm and arteriovenous malformations,and take part in hybrid operation.
Sampling Method: Non-Probability Sample
Enrollment: 556 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Changes in hemorrhage event rate from the beginning of surgery to 48 hours after surgery | From the beginning of surgery to 48 hours after surgery
  Hemorrhage event include intracranial hemorrhage caused by non-surgical reasons, as well as other organs or parts of the massive bleeding or small bleeding, Including subperitoneal hemorrhage, intraocular hemorrhage, gross hematuria, epistaxis time prolonged or repeated, gastrointestinal bleeding, hemoptysis, subconjunctival hemorrhage, hematoma greater than 5cm, bleeding difficult to control the and so on.

SECONDARY OUTCOMES:
Changes in ischemia event rate from the beginning of surgery to 48 hours after surgery | From the beginning of surgery to 48 hours after surgery
  Ischemia event include Cerebral infarction and transient ischemic attack.
Intraoperative blood loss | During the surgery
  All the blood lost during the surgery should be collected and measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No